CLINICAL TRIAL: NCT06332625
Title: The Fingerprinting of Inherited Leukoencephalopathies: A New Brain Imaging, Genetic and Clinical Assessment (FIABA)
Brief Title: The Fingerprinting of Inherited Leukoencephalopathies: A New Brain Imaging, Genetic and Clinical Assessment
Acronym: FIABA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Oasi Research Institute-IRCCS (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); IRCCS Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: PNRR-MR1-2022-12375648
Record Dates: First submitted 2024-02-23; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Leukoencephalopathies
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Brain quantitative magnetic resonance imaging — Identification and predictability of early structural and metabolic markers from 3T and 7T quantitative magnetic resonance imaging (qMRI)

SUMMARY:
Inherited leukoencephalopathies are a broad spectrum of genetically determined disorders, characterized by specific involvement of the white matter of the central nervous system. These pathologies are almost as common as other acquired white matter disorders, such as acute disseminated encephalomyelitis and multiple sclerosis. The onset can occur at any age, from prenatal life to adulthood, and the clinical picture is mostly progressive, but can also be non-evolving or, rarely, improve over time. Thanks to new diagnostic approaches, including next-generation genetic sequencing and recognition of magnetic resonance imaging patterns, in recent years the investigators have witnessed a significant increase in the number of genetically defined leukoencephalopathies. However, despite advances in genetic studies, inherited leukoencephalopathies include a large number of inherited white matter diseases in children and adults and remain of unknown cause in many patients (about 40%). This significant percentage of cases of unknown etiology represents a major challenge for public health, both in prognostic terms and, consequently, economically. However, even in leukoencephalopathies of genetically determined cause, the absence of specific biomarkers can be a limiting factor in the design and execution of clinical studies in search of promising therapies. As in other fields of neurology, the integration of clinical and genetic data with brain MRI data plays a fundamental role in the diagnostics of subjects affected by these pathologies. Currently, the methodologies commonly used in magnetic resonance imaging are qualitative, and evaluate brain lesions through the contrast between white and gray matter. The lack of specific biomarkers is therefore a limiting factor in the design of therapeutic challenges. In this regard, the development of new multiparametric quantitative magnetic resonance imaging (qMRI) methods could allow the investigators to identify new biomarkers to assess the etiology behind leukodystrophies, increasing diagnostic power and understanding the progression or improvement of leukoencephalopathy for both future trials and existing therapies. In this perspective, recent rapid "transient-state" magnetic resonance imaging methods, such as MR Fingerprinting (MRF), have proven effective in efficiently separating different components of brain tissue. These techniques consist of rapid and highly undersampled acquisitions performed by continuously changing the MR sequence parameters, thus obtaining a signal evolution that is unique for each combination of underlying tissue properties. Furthermore, if these techniques have already shown their validity at 3 Tesla, they could be even more informative in 7T MRI where the use of qMRI could provide more details thanks to the high image resolution.

The project's objective is to evaluate and validate new and innovative quantitative magnetic resonance imaging (qMRI) methodologies at both clinical and ultra-high fields in inherited leukodystrophies and those of unknown etiology.

This is a national, multi-institutional, multicenter exploratory study on the potential identification and predictability of early structural and metabolic markers in quantitative MRI at 3T and 7T in the diagnosis and follow-up of leukodystrophy and leukoencephalopathy in adults and during development.

The study will include multiple sub-studies:

1. A cross-sectional study in leukoencephalopathies at clinical fields.
2. A longitudinal study in leukoencephalopathies at 3T: natural history and therapy outcomes.
3. A cross-sectional and longitudinal study at 7T: The added value of ultra-high-field Magnetic Resonance Imaging in leukoencephalopathies.

ELIGIBILITY:
Inclusion Criteria:

* For MRI examinations at clinical fields:

  * Patients under 30 years of age with leukoencephalopathy already diagnosed and listed in institutional clinical databases or arriving at any Operational Unit during the project that meet the standard inclusion criteria;
  * Typical development patients under 30 years of age undergoing brain MRI for clinical reasons other than leukoencephalopathy (e.g., headache) with normal brain MRI results.
* For ultra-high field MRI (7T) examination:

  * Patients with leukoencephalopathy aged between 8 and 30 years, who are capable of cooperating with an MRI examination.
  * Patients suffering from leukoencephalopathy, who have already undergone a clinical field MRI (≤3T) as part of their diagnostic or research clinical pathway according to the diagnostic flowchart identified and shared with other institutes, and who present inconsistencies between clinical and imaging profiles or white matter patterns on clinical field imaging.

Exclusion Criteria:

* All subjects with absolute contraindications to undergoing an MRI exam, as determined by the medical history questionnaire.
* Patients with severe clinical conditions, such as the presence of a tracheostomy.

Additionally, further exclusion criteria for subjects participating in the 7T study will include:

* Age under 8 years;
* Inability to cooperate with undergoing an MRI exam.

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 100 subjects with leukoencephalopathy will undergo quantitative analysis at clinical field strengths, of which 20 will also be subjected to 7T MRI.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2025-11-22 (Estimated)

PRIMARY OUTCOMES:
Quantitative Susceptibilty Mapping, QSM | every year for two years
  The Relative magnetic susceptibility values (in units of parts per billions [ppb], with respect to water magnetic susceptibility) registered in subcortical structures and nuclei
Fractional Anisotropy, FA | every year for two years
  FA values (a fractional number between 0 and 1), registered in lesioned white matter and normal-appearance white matter
Mean Diffusivity, MD | every year for two years
  MD values (in units of square millimeters per second [mm²/s]), registered in lesioned white matter and normal-appearance white matter
Relaxation times | every year for two years
  Values of longitudinal (T1) and transverse (T2) relaxation times (in units of milliseconds [ms]), registered in grey matter, lesioned white matter, normal-appearance white matter, and subcortical nuclei
Myelin water fraction, MWF | every year for two years
  MWF values (a fractional number between 0 and 1), registered in grey matter, lesioned white matter, normal-appearance white matter, and subcortical nuclei
Neuromotor skills | every year for two years
  Gross Motor Function Classification System (GMFCS) is a motor scale that categorizes patients' motor skills into 5 levels. Each level corresponds to a range of motor functions, with Level 1 representing mild symptoms and Level 5 being the most severe
Neuromotor skills | every year for two years
  Movement Disorders-Childhood Rating Scale Revised (MD-CRS R) has a score ranging from 0 and 100 with deficits below 70

SECONDARY OUTCOMES:
Epilepsy symptoms | every year for two years
  The presence of epilepsy symptoms (presence or absence)
Electroencephalography features | every year for two years
  Electroencephalography alteration (EEG-alteration) (presence or absence)
Neuro-psychological profile | every year for two years
  Wechsler Intelligence Scale for Children (WISC) has a score ranging from 0 and 100 with deficits below 70

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Associazione Oasi Maria SS Troina, Troina, Enna
  - Ospedale San Raffaele, Milan
  - Fondazione Istituto Neurologico Carlo Besta, Milan

IPD SHARING:
Plan to Share IPD: No